CLINICAL TRIAL: NCT06724523
Title: Pre- and Post- Descriptive Data of Language Outcomes in Deaf Children
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 478856; R21DC021024 (NIH)
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Sign Language Skills
Keywords: sign language; deaf; instruction
MeSH Terms: conditions — Sign Language

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Deaf children: Deaf children attending deaf education programs
  Interventions: Behavioral: Business-as-usual instruction

INTERVENTIONS:
Behavioral: Business-as-usual instruction — Deaf children are receiving business-as-usual instruction in sign language in deaf education programs.

SUMMARY:
Deaf children between ages of 4-10 will provide pre and post data by responding to three prompts in sign language and written language at the beginning and end of a year. This data will provide information on the developmental trends and characteristics of deaf children who will receive SISI the following year.

ELIGIBILITY:
Inclusion Criteria:

* Deaf children between 4 and 10 years old attending deaf education programs

Exclusion Criteria:

* Non-deaf children

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Deaf children between 4 and 10 years old attending deaf education programs
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Sign Language Skills | From enrollment to the end of treatment 9 academic months later.
  Deaf children's sign language skills will be evaluated.

SECONDARY OUTCOMES:
Written Language Skills | From enrollment to the end of treatment 9 academic months later.
  Deaf children's written language skills will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee, Knoxville, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Under a data-sharing agreement that is in compliance with the internal policy at UTK, non-identifying data can be shared with other researchers for a minimum of 10 years on the University of Tennessee Research and Creative Exchange (TRACE). The raw data consists of videos of teachers, which will not be shared to maintain confidentiality. The processed data will be in the form of percentages for individual teachers across an academic year documented in a .csv file (Excel). Center for Open Science Foundation (OSF) is a free and open source project management tool that supports researchers throughout their entire project lifecycle. OSF also allows people to locate this data through project names, author names, and study keywords.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: December, 2026 to December, 2036
Access Criteria: Researchers may contact the principal investigator for additional supporting information not available on OSF.